CLINICAL TRIAL: NCT01391624
Title: Study on the Possible Effects of Diet Supplementation With Essential Fatty Acids in Chocolate Craving Volunteers
Acronym: OMEGA3CHOCO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: José Carlos Fernandes Galduróz, MD, PhD, Adjunct Professor in the Department of Psychobiology of the Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Omega3-chocolate-001
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Addictive Behavior; Abstinence Syndrome
Keywords: chocolate; craving; addiction; compulsion
MeSH Terms: conditions — Behavior, Addictive; Compulsive Behavior | interventions — Linseed Oil; Fatty Acids, Essential; Paraffin; 2-(2-(2-chloro-3-(2-(3,3-dimethyl-5-sulfo-1-(4-sulfo-butyl)-3H-indol-2-yl)-vinyl)-cyclohex-2-enylidene)-ethylidene)-3,3-dimethyl-1-(4-sulfo-butyl)-2,3-dihydro-1H-indole-5-carboxylic acid; Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega 3 (Experimental): The group was treated with omega 3 fatty acids for 2 months.
  Interventions: Drug: Flaxseed oil
- Placebo (Placebo Comparator): The group received paraffin with dye in order to mimic the visual aspects of omega 3 fatty acid capsules.
  Interventions: Drug: Paraffin + # 2 dye

INTERVENTIONS:
Drug: Flaxseed oil — 3 g (3 capsules/day) of flax oil for a period of 8 weeks
  Other Names: DHA; EPA; Essential fatty acids
  Arms: Omega 3
Drug: Paraffin + # 2 dye — 3 capsules of mineral oil (ineffective) for 8 weeks.
  Other Names: Mineral oil
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether essential polyunsaturated acids (omega 3) are capable of reducing chocolate craving symptoms in healthy patients.

Our hypothesis is that the omega 3 fatty acids have properties which stabilize and normalize neuronal functioning in many conditions, including chocolate craving.

DETAILED DESCRIPTION:
Polyunsaturated fatty acids (of the omega 3 subtype) are fundamental in human diet, as they are components of cellular membranes, guaranteeing their fluidity and their functions of separating intracellular and extracellular means and transporting several substances to and from cellular microenvironment.

Modern theories profess that lack of omega 3 fatty acids in western diets may be the cause of several deletery changes in neuronal physiology, which may cause or make worse several pathological conditions, such as depression, mood instability, and drug craving. The role of serotonin as the main lacking component in the conditions is well documented, and it is thought that omega 3 is important in the synthesis, transportation, and ultimately the activity of this neurotransmitter.

Out theory states that supplementation with these acids can restore normal neuron balance, improving the condition of chocolate craving patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chocolate compulsion or craving, ECAP score > 12.

Exclusion Criteria:

* Psychiatric disease of any sort (by the DSM IV criteria, Use of psychoactive drugs of any sort, BMI > 25 (kg/m2).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes in the MBES score (used to quantify chocolate compulsion) from baseline. | 2 months after enrollment
  The MBES is an objective scale used to quantify compulsion and classify chocolate cravers in three categories: low, moderate and severe cravers. The scale was applied to all volunteers at baseline and 2 months after enrollment in the study, and comparisons were made to establish if there was efficacy of treatment with omega 3 when compared with placebo (with decreased grades in the MBES scale).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Prior, Student, Study Chair — Student
Locations (1):
- Universidade Federal de São Paulo (Federal University of São Paulo); Departamento de Psicobiologia (Department of Psychobiology), São Paulo, São Paulo, Brazil